| | 1 |
|---|---|
| | 2 |
| | 3 |
| | 4 |
| | 5 |
| | 6 |
| | 7 |
| | 8 |
| | 9 |
| 1 | 0 |
| 1 | 1 |
| 1 | 2 |
| 1 | 3 |

15

# Clozapine OpTimal Timing for Optimal moNitoring and Side effects (COTTONS)

(November 2024)

# PROTOCOL TITLE 'Clozapine OpTimal Timing for Optimal moNitoring'

| Protocol ID | COTTONS |
|---|---|
| Short title | Clozapine OpTimal Timing for Optimal moNitoring and Side effects |
| EudraCT number | n.a. |
| Version | 2.0 |
| Date | 22 November 24 |
| Coordinating investigator | A. Abdul Roda, MSc |
| | E-mail: a.abdulroda@amsterdamumc.nl |
| | Phone: +31(0)617789903 |
| Co-investigators | Participating sites: |
| | GGZ NHN, Alkmaar |
| | - L. Kaya, MD |
| | - M. Musters, MD |
| | Noordwest ziekenhuisgroep, Alkmaar |
| | - F. Ph. Mulder, PharmD |
| | - E. ten Boekel, PhD |
| | - Dr. S. Simsek, MD, PhD |
| | - R. Fijn, PharmD, PhD |
| | Albert Schweitzer ziekenhuis, Dordrecht |
| | M.M. Beex-Oosterhuis, PharmD, PhD |
| | University Medical Center Groningen, Groningen |
| | prof. D.J. Touw, PharmD, PhD |
| Principal investigator(s) (in | Noordwest ziekenhuisgroep, Alkmaar |
| Dutch: hoofdonderzoeker/<br>uitvoerder) | P.C.D. Bank, PharmD, PhD |
| | Email: <u>pcd.bank@nwz.nl</u> |
| | Phone: 088 085 5110 |
| | GGZ Noord-Holland-Noord |
| | S.R.T. Veerman, MD, PhD |
| | Email: <u>s.veerman@ggz-nhn.nl</u> |
| | Amsterdam UMC, locatie AMC |
| | Prof. R.A.A. Mathôt, PharmD, PhD |

| | Email: r.mathot@amsterdamumc.nl |
|---|---|
| | Phone: 020 566 3327 |
| Sponsor (in Dutch: verrichter/opdrachtgever) | GGZ NHN |
| Subsidising party | N.A. |
| Independent expert (s) | N.A. |
| Laboratory sites | NWZ Alkmaar |
| | Juliana van Stolberglaan 13, 1814 HB Alkmaar |
| | 072 548 4444 |
| Pharmacy | N/A |

# PROTOCOL SIGNATURE SHEET

| Name | Signature | Date |
|---|---|---|
| Sponsor: | | |
| GGZ NHN | | 18-11-2024 |
| S.R.T. Veerman, MD, PhD<br>psychiatrist GGZ NHN<br>board member Dutch Clozapine<br>Collaboration Group | | |
| Principal Investigator: | | |
| P.C.D. Bank, PharmD, PhD hospital pharmacist & clinical pharmacologist, co-chair clinical pharmaceutical laboratory, North West Clinics Member Dutch Clozapine Collaboration Group | | 18-11-2024 |
| Prof. R.A.A. Mathôt, PharmD, PhD<br>hospital pharmacist &<br>clinical pharmacologist,<br>Amsterdam UMC, location AMC | | |

| 21<br>22<br>23 | TABLE OF CONTENTS | |
|---|---|---|
| 24 | INTRODUCTION AND RATIONALE | 8OBJECTIVES |
| 25 | | 13STUDY DESIGN |
| 26 | | 14STUDY POPULATION |
| 27 | | 15Population (base) |
| 28 | | 15Inclusion criteria |
| 29 | | 15Exclusion criteria |
| 30 | | 15Sample size calculation |
| 31 | | 15TREATMENT OF SUBJECTS |
| 32 | | 16INVESTIGATIONAL PRODUCT |
| 33 | | 16NON-INVESTIGATIONAL PRODUCT |
| 34 | | 16METHODS |
| 35 | | 17Study parameters/endpoints |
| 36 | | 17Main study parameter/endpoint |
| 37 | | 17Secondary study parameters/endpoints |
| 38 | | 17Other study parameters |
| 39 | | 18Randomisation, blinding and treatment allocation |
| 40 | | 18Study procedures |
| 41 | | 18Withdrawal of individual subjects |
| 42 | | 18Specific criteria for withdrawal (if applicable) |
| 43 | | 18Replacement of individual subjects after withdrawal |
| 44 | | 18Follow-up of subjects withdrawn from treatment |
| 45 | | 18Premature termination of the study |
| 46 | | 18SAFETY REPORTING |
| 47 | | 19STATISTICAL ANALYSIS |
| 48 | | 20Primary study parameter(s) |
| 49 | | 20Secondary study parameter(s) |
| 50 | | 22Other study parameters |
| 51 | | 23Interim analysis (if applicable) |
| 52 | | 23ETHICAL CONSIDERATIONS |
| 53 | | 24Regulation statement |
| 54 | | 24Recruitment and consent |
| 55 | 24Obje | ection by minors or incapacitated subjects (if applicable) |
| 56 | | 24Benefits and risks assessment, group relatedness |
| 57 | | 24Compensation for injury |
| 58 | | 24Incentives (if applicable) |
| 59 | 24ADMINISTF | RATIVE ASPECTS, MONITORING AND PUBLICATION |
| 60 | | 25Handling and storage of data and documents |
| 61 | | 25Monitoring and Quality Assurance |
| 62 | | 26Amendments |

| 26Annual progress report | 63 |
|--------------------------------------------------------|----|
| 26Temporary halt and (prematurely) end of study report | 64 |
| 26Public disclosure and publication policy | 65 |
| 26STRUCTURED RISK ANALYSIS | 66 |
| 26TIME SCHEDULE | 67 |
| 26REFERENCES | 68 |
| 27 | 69 |
| | 70 |

#### LIST OF ABBREVIATIONS AND RELEVANT DEFINITIONS

71 72

ABR General Assessment and Registration form (ABR form), the

application form that is required for submission to the accredited Ethics Committee; in Dutch: Algemeen Beoordelings- en Registratieformulier (ABR-formulier)

AUC Area Under the Curve

CI Clearance

Cmax Maximum Concentration
CV Coefficient of Variation
EHR Electronic Health Record
GCP Good Clinical Practice

GDPR General Data Protection Regulation; in Dutch: Algemene

**Verordening Gegevensbescherming (AVG)** 

IC Informed Consent

ICC Class Correlation Coefficient

IIV Interindividual Variability (synonyms are interpatient of

between-patient variability)

IOV Interoccasion Variability (synonyms are intrapatient of

within-patient variability)

Ke The elimination rate constant, is the fraction of a drug that

is eliminated from the body over a set unit of time

MIPD Model-Informed Precision Dosing
NONMEM Nonlinear Mixed-Effects Modelling
PANSS Positive and Negative Syndrome Scale

PD Pharmacodynamics
PE Prediction Error
PK Pharmacokinetics

PopPK Population pharmacokinetics
RMSE Root Mean Square Error

SPC Summary of Product Characteristics; in Dutch: officiële

productinformatie IB1-tekst

Sponsor The sponsor is the party that commissions the

organisation or performance of the research, for example a pharmaceutical company, academic hospital, scientific organisation or investigator. A party that provides funding for a study but does not commission it is not regarded as the sponsor, but referred to as a subsidising party.

Equilibrium where drug intake equals elimination,

maintaining constant average concentration (= approx. 4-5x

the half-life).

T<sub>1/2</sub> Half-life, time it takes for the concentration to be halved

TDM Therapeutic Drug Monitoring

Therapeutic window Range of plasma drug concentrations spanning the

minimum concentration for clinical efficacy and toxicity

Tmax Time to Maximum concentration

Trough Lowest concentration of a drug in the bloodstream, usually

iust before intake of the next dose

UAVG Dutch Act on Implementation of the General Data

Protection Regulation; in Dutch: Uitvoeringswet AVG

Vd Distribution of volume

WMO Medical Research Involving Human Subjects Act; in Dutch:

Wet Medisch-wetenschappelijk Onderzoek met Mensen

Steady state

#### **SUMMARY**

#### Rationale:

Therapeutic drug monitoring (TDM) is essential for clozapine and can enhance therapeutic outcomes and minimize side effects. As of yet, research on (nor)clozapine concentrations and their association to metabolic side effects is limited and inconclusive. Unfortunately, not enough is known about individual risk factors for developing metabolic side effects to personalize clozapine treatment. It would be desirable to have another way to predict which clozapine users are at increased risk of developing severe side effects. Current guidelines are based on limited evidence, potentially resulting in inconsistent or suboptimal monitoring and management.

#### **Objective:**

The primary objective is to evaluate the correlation between (nor)clozapine kinetics and serum level HbA1c. Secondary objectives include validating an existing population pharmacokinetic model, assessing the validity of the current 12-hour post-intake sampling practice, determining the optimal sampling window for once-daily clozapine TDM and assessing the correlation of other metabolic and multiple laboratory parameters and influence of demographic and clinical parameters on the pharmacokinetics and -dynamics of clozapine and norclozapine.

#### Study design:

This is a non-interventional single-center cohort study involving prospective data collection for the primary (pharmacodynamic) analysis. This will be supplemented with retrospective population pharmacokinetic analyses. Using pharmacokinetic/pharmacodynamic modelling and statistical analysis will be used to evaluate the relation to side effects as well as optimize the sampling time for clozapine. Demographic, clinical and laboratory data are collected routinely based on current standard practice.

#### Study population:

The study includes patients (18-70 years) diagnosed with treatment-resistant schizophrenia or schizoaffective disorder who are on a registered, stable dose of clozapine. Participants must have a known smoking status and have their times of intake and sampling registered. To ensure comparability of (nor)clozapine concentrations, pregnant women will be excluded as well as plasma levels affected by acute inflammation/infection/intoxication and/or cessation or dose change of interacting co-medication or tobacco containing products seven days prior to sampling. Clinical parameters such as baseline severity of illness, duration of illness and duration of clozapine treatment will be assessed to describe the study population.

#### Main study parameter/endpoint:

The main study parameter is to evaluate the correlation between (nor)clozapine kinetics and serum level HbA1c. The correlation between (nor)clozapine concentrations and ratio and HbA1c will be assessed using a PK-PD turn over model.

# Nature and extent of the burden and risks associated with participation, benefit and group relatedness.

Not applicable for this retrospective non-interventional study.

#### INTRODUCTION AND RATIONALE

# Background clozapine

121 122 123

124

125

126

127 128

129 130

131

132133

134

135

136

137 138

139

140

141

142

143

144

145 146

147

148149

150

151

152

153 154

155

156 157

158 159

160 161

162

163 164

165 166

167

168

169 170

171 172

173174

Clozapine has proven to be superior to other antipsychotics in treatment of refractory schizophrenia. Therapeutic drug monitoring (TDM) is strongly recommended for clozapine, a relatively well-studied compound among antipsychotics. As clozapine levels show large interand intraindividual variation, TDM helps to increase efficacy and reduce prevalence of side effects and toxicity (1-4). A systematic review and meta-analysis has shown a higher risk of non-response in the treatment of refractory schizophrenia or schizoaffective disorder when plasma levels are below the threshold of 350 to 400 µg/l. Other publications have shown that increased plasma levels (> 750 µg/L) are associated with anticholinergic side effects and the occurrence of seizures (4). Clozapine is known to cause more serious metabolic side effects than other antipsychotics (5). Up to 80% of the patients are overweight and 45 to 58% have metabolic syndrome, while hyperglycemia and hypertension are often undertreated. Cardiometabolic disorders are therefore the most common cause of premature death in schizophrenia. Clozapine-induced agranulocytosis (CIA) is much rarer, occurring in 0.4% of clozapine users and the risk of death is 10% (6). Nevertheless, fear of CIA is often a reason not to choose clozapine. Norclozapine, clozapine's main metabolite, may contribute to some extent to the therapeutic effect and side effects of clozapine. Though, its precise role is yet inconclusive (7-10). Due to its unknown clinical relevance, many laboratories do not measure norclozapine. It is likely that norclozapine, due to its stronger effect as an inverse agonist on the serotonin 5-HT2C receptor, causes weight gain and metabolic abnormalities, which are associated with a lower quality of life and somatic comorbidities such as diabetes mellitus type II, cardiovascular diseases and higher mortality (7). This is further supported by other small studies where norclozapine caused insulin resistance in animals(11), an association between norclozapine levels and elevated triglycerides, elevated cholesterol, and weight gain (12) was found or with a higher waist circumference and higher HbA1c (8). Studies with either CYP1A2 induction through smoking (8) or inhibition through fluvoxamine (13) show norclozapine concentrations to be associated with waist circumference, HbA1c, and body mass index (BMI) (8) or a lower weight and metabolic parameters (insulin, glucose and triglycerides) (8, 13, 14). Finally, two studies contradict this association as a clozapine/norclozapine ratio > 2 appears to be most beneficial regarding cardiometabolic outcomes according to Polcwiartek et al. (15), whereas Lu et al. could not confirm this at a ratio of 3.7 (14). Regarding the level of granulocytes, only one study has shown a higher norclozapine concentration to be more beneficial than a higher clozapine concentration after long-term use of clozapine (16). As of yet, research on (nor)clozapine concentrations and their association to metabolic side effects is limited and inconclusive. For both patients and healthcare providers, blood tests and fear of side effects are the main reasons to postpone or even abandon clozapine treatment (17). Unfortunately, not enough is known about individual risk factors for developing metabolic side effects to truly personalize clozapine treatment. It would be desirable to have another way to predict which clozapine users are at increased risk of developing severe side effects. Because of this, current guidelines differ in their advice regarding metabolic screening.

#### Therapeutic drug monitoring of clozapine

Based on the information mentioned above, the recommended window for therapeutic drug monitoring for clozapine is  $350\text{-}700~\mu\text{g/L}$  for both once- and twice-daily dosing. Some patients respond well on lower or higher levels; the latter is acceptable as long as higher levels are tolerable. The therapeutic window is based on trough concentrations (i.e., approximately 12 hours after the evening dose) from studies using a divided dosing regimen(18, 19). Similar to twice-daily dosing, current practice for once-daily dosing of clozapine advises a sample to be collected at least 12 hours after intake or within a window of 10-14 hours after intake. It is however unknown if the concentration-effect relations of once- and twice-daily dosing are similar. Additionally, clinical laboratories do not have a

uniform general practice regarding sampling times, resulting in variability in preferred sampling times and windows (1, 3, 4, 20).

As of yet, while often used in daily practice, there is no conclusive evidence as to the adequacy and suitability of this sampling time for once-daily dosing. Clozapine's pharmacokinetic properties further question this suitability. It has a biphasic elimination with a mean elimination half-life of 12-16 hours (3). The range is 6-26 hours, which after a single dosage of 75 mg was reported to be 7.9 hours that increased to 14.2 hours after reaching steady state (after one week) (21). Theoretically, a mean half-life of 12 hours and sampling time of 12 hours could lead to inadequate and inconsistent samples. This might be suitable for twice-daily dosing, where a 12-hour sample would be a trough, but this might not be the case for once-daily dosing. With once-daily dosing concentrations at 12 hours after ingestion may be adequate (within the therapeutic window) but subtherapeutic after 24 hours. Furthermore, smoking influences the metabolism such that a shorter half-life is reported (21).

#### Pharmacokinetics of clozapine in relation to dosing

177

178179

180

181 182

183 184

185

186 187

188 189

190

191 192

193

194

195

196

197

198 199

200

201

202203

204

205

206

207208

209

210211

212213

214215

216

217218

219

220221

222

223

224

225226

227

228

One way to understand the pharmacokinetic variability of such compounds and provide individualised treatment strategies is by using population pharmacokinetics (popPK) models. These serve as useful tools within the framework of the model-informed precision dosing (MIPD). A previous study determined the comparability of once- and twice-daily dosing based on popPK analyses as well as the effect of once-daily dosing on clozapine and norclozapine concentrations (22). Their simulations show a 30% higher 12 hr-post dose concentration with once-daily (400 mg) dosing versus twice-daily (2x 200mg) dosing and a 30% lower trough (24 hr-post dose) when dosed once-daily compared to twice-daily. A higher once-daily dosage, 700 mg, shows 12 hr-post dose concentrations to lie above the upper limit and a trough (24 hr-post dose concentration) to be within the therapeutic window but almost half the 12 hr-post dose concentration (788 µg/L vs 425 µg/L). This suggests the current sampling time of 12 hr-post dose to be inadequate for once-daily dosing. This is further supported by Procyshyn et al. as well as Zwaag et al. who noted simulated 12 hr-post dose concentrations to be 23% higher after a single evening dose versus twice-daily dosing (23, 24). Neither of these two studies included norclozapine in their assessment. This in contrast to the study by Kitagawa et al. where no significant differences were found in estimated peak and trough samples of clozapine and norclozapine dosed once-versus twice-daily (400 mg/day) (25). The Dutch Clozapine Working group recommends increasing the lower limit of clozapine's therapeutic range by 23% for 12-hr post evening dose samples in patients with once-daily dosing based on the study by Zwaag et al (4, 23).

For a valid interpretation of the clozapine/norclozapine ratio, the clozapine dosage regimen, and blood sampling interval are important. Sources of large variability in pharmacokinetics of clozapine that affect CYP1A2 metabolism are smoking behaviour (polycyclic aromatic hydrocarbons in cigarette smoke induce CYP1A2), caffeine consumption (CYP1A2) substrate), and estrogen and progesterone levels (inhibit CYP1A2). Excessive smoking is correlated with reduced plasma levels of both CLO and NCLO. Coffee consumption is correlated with increased CLO and NCLO plasma levels and negatively correlated with the CLO/NCLO plasma level ratio. In premenopausal women CLO levels are higher compared to postmenopausal women (26). Pharmacokinetic drug-drug interactions are caused by the inhibition or induction of CYPs. Fluvoxamine increases the CLO/NCLO ratio through inhibition of the CYP1A2 enzyme. The demethylation of CLO to NCLO is reduced, resulting in an increase of the CLO plasma level and decrease of the NCLO plasma level (26). Pro-inflammatory cytokines interleukin (IL)-6 and IL-1 inhibit CYP1A2, which can be detected indirectly using the biomarker C-Reactive Protein (CRP). Furthermore, CLO is highly bound to the acute phase protein alpha-1-acid glycoprotein (AGP) and less to serum albumin (95% of CLO binds to AGP). During inflammation, concentrations of AGP increase, resulting in a decreased CLO unbound fraction. Pharmacogenetics of the also affects pharmacokinetics of clozapine. For example, asian ancestry is associated with lower CYP1A2 activity compared to other ethnic groups. Additionaly, genetics may also account for variability in response tot

clozapine. It is reported that transcriptional activity of the M1 receptor gene is correlated with anticholinergic burden (26).

Finally, CLO clearance is affected by age, sex, ethnicity, and smoking status. Higher age results in a reduction in CLO clearance for both male and female smokers and non-smokers of all ethnicities. Females have decreased CLO clearance compared to males. Patients of Afro-Caribbean ethnicity have increased CLO clearance, whereas patients of Asian ethnicity have decreased CLO clearance compared to their White counterparts. Additionally, smokers have increased CLO clearance compared to non-smokers (26).

In addition to the CLO/NCLO ratio additional biomarkers to predict the CYP1A2 activity could be useful in clinical practice. Pu et al have reported that in rats the ratio of the concentrations of the amino acids phenylalanine and tyrosine in serum is highly correlated with the expression of the CYP1A2 gene and the activity of the CYP1A2 enzyme. This biomarker could be useful in prediction of the clearance of clozapine by this enzyme (27).

#### Pharmacokinetic modelling

231232

233

234

235

236

237238

239240

241

242243

244

245 246

247

248

249

250

251

252

253254

255

256257

258259

260

261262

263

264 265

266267

268

269

270

271272273

274

275

276

277278

279

280

281 282

283

Population PK models may be used to determine the sampling time or window that yields the most precise estimation of pharmacokinetic parameters through simulations and optimization techniques. Since several models have been developed for clozapine, a careful selection based on suitability is applied. In this case, a valid popPK model should be developed including Dutch patients, once-daily dosing regimen, trough samples of both clozapine and norclozapine (up until 24 hours after ingestion) and include sufficient information during the elimination phase. Geers et al. describes a popPK model for clozapine based on Dutch patients. However, this model only included samples of patients who are dosed twice-daily, fewer samples were taken between 8-24 hours after intake (and thus during the elimination phase) and their model was based on two-time point sampling strategies for AUC (28). Perera et al. studied optimal sampling points through modeling, but did so for twice-daily dosing regimen based on AUC based monitoring as well and concluded three-time point strategies. They also concluded that trough concentrations show an excellent correlation to exposure (29). Geers et al. concluded the same for twice-daily dosing regimen (AUC0-12) (28). Shang et al. used population PK/PD modeling to study the relationship between exposure of clozapine (AUC) and the Positive and Negative Syndrome Scale (PANSS) (30). They found the AUC to be a better predictor as PANSS score showed little relationship with trough concentrations of clozapine. However they mention that this is probably due to the slow onset of antischizophrenic effect after reaching steady state. Furthermore they only included Chinese patients with a twice-daily dosing regimen. In addition none of these models included norclozapine. The recent model by Beex et al. is based on Dutch patients, trough samples of both clozapine and norclozapine as well as once- and twice-daily dosing regimen (22). They mention model misspecification in the absorption phase. This might be due to the occurrence of a first-pass effect and could have been described if more samples had been taken during the absorption phase. However, this should not be relevant to this study which focuses on sampling times during the elimination phase. Therefore this model is most suitable to be used to study and find the optimal sampling time or window. Its suitability will be further examined by performance of an external validation.

#### Pharmacokinetics/pharmacodynamics and metabolic side effects

Metabolic side effects of clozapine comprise weight gain, dyslipidemia and hyperglycemia, which can result in a metabolic syndrome, associated with an increased risk for type 2 diabetes mellitus and cardiovascular disease (5). NCZ is hypothesised due to its stronger action as an inverse agonist on the serotonin 5-HT2C receptor to cause weight gain and metabolic changes, which are associated with a lower quality of life, somatic comorbidity, and a higher mortality (7).

In a small low-quality meta-analysis (n=120) a positive correlation was found between clozapine concentrations and elevated triglycerides, heart rate, and overall combined adverse drug reaction (12). Furthermore, a positive correlation was found between norclozapine plasma levels and triglycerides, cholesterol, and weight gain. In short, at

present there is too little evidence to identify the role of the clozapine/norclozapine plasma level ratio in the minimisation of clozapine side effects. In addition, the correlation of CLO(&CNLO) concentration with metabolic markers might be affected by cortisol and genetics of the glucocorticoid receptor (31). Finally, other genetic markers known to modulate the basic risk of metabolic syndrome might play a role in this correlation between the correlation of the CLO(&CNLO) concentration and the increase in metabolic markers (32).

#### Personalised clozapine treatment

Since clozapine is mostly given to patients with treatment-resistant schizophrenia, a clear defined sample time is required in order to interpret their plasma concentrations and optimize their treatment through TDM. Inadequate interpretation may lead to suboptimal treatment efficacy or increased risk of adverse effects. Furthermore the relation of adverse effects, especially metabolic and granulocyte, to (nor)clozapine concentration has yet to be researched well in order to improve screening and optimize treatment. Based on earlier studies it is suggested that current sample times may fit a twice-daily dosing schedule and not a once-daily dosing schedule. Thus in this study the difference between the (nor)clozapine concentrations at 12-hours post intake and the concentration at other time points within the 10-14 hours sampling window will be evaluated for once-daily dosed clozapine. To this end, the model by Beex et al. will be validated with independent data. Through predicted concentrations, we aim to contribute novel insights into the optimal timing of sample collection as well as insight into the development of metabolic and granulocyte side effects, addressing the existing knowledge gap and enhancing the precision of therapeutic drug monitoring in this population.

This research will not only provide more knowledge about risk factors for developing general side effects of clozapine, metabolic side effects, constipation, and chronic neutropenia, but will also improve metabolic screening in clozapine users through better implementation of metabolic screening.

Version number: 2, 22-11-2024

#### **OBJECTIVES**

315 316 317

#### Primary Objective:

318

# 319

# 320

#### 321 322 323 324

325 326 327

328 329 330

332 333 334

331

335 336 337

338 339

340 341 342

351 352 353

354

355

356 357 358

359

#### To evaluate the correlation of (nor)clozapine kinetics and serum level HbA1c

- Secondary Objectives: To validate an existing population model with independent data.
  - To study the validity of current practice (12-hr post intake) sampling times within a window of 4 hours (10-14 hours post intake) for TDM of once daily dosed clozapine
  - To identify the optimal sampling time or window for TDM of clozapine based on predicted concentration-time profiles up until 24-hours post intake.
  - To investigate the influence of the following covariates on the pharmacokinetics of clozapine, the metabolite norclozapine (and CZ/NCZ ratio):
    - 0 age
    - estradiol (indirectly through demographic data [premenopausal or postmenopausal female / male).
    - comedication with fluvoxamine (dosage) and other medication
    - ethnicity (Asian ancestry is associated with lower CYP1A2 activity compared to other ethnic groups).
    - pharmacogenetics of the metabolic enzymes CYP2C19 and CYP3A4
    - smoking behaviour (yes/no and amount)
    - inflammation markers (C-reactive protein (CRP) and Erythrocyte Sedimentation (BSE))
    - phenylalanine and tyrosine (a higher ratio of phenylanlanine/tyrosine is associated with a higher CYP1A2 activity) (27).
  - To evaluate the correlation of (nor)clozapine concentrations and/or ratio on:
    - Other metabolic parameters such as: fasting glucose, insulin, HOMA-IR, triglycerides, HDL, LDL, total cholesterol, BMI, abdominal circumference, blood pressure and heart rate.
    - Absolute neutrophil count (ANC) and total white cell count (TWC).
    - General side effects of clozapine using the Glasgow Antipsychotic Side-effect Scale for Clozapine (GASS-C) (33).
    - Defecation frequency per week and consistency using the Bristol Stool Form Scale (BSFS).
    - Positive and Negative Syndrome Scale (PANSS-6), regarding severity of schizophrenia
  - To evaluate the effect of cortisol concentration and genetics of known relevant loci related on the correlation of (nor)clozapine concentrations and/or ratio on the metabolic markers (31,32)

#### STUDY DESIGN

This is a (non-interventional) single-center cohort study. (Out)patient data will be collected from the mental healthcare organization GGZ-NHN and the laboratory of NorthWest clinics. For all endpoints a baseline value is required. The inclusion period will start 01-12-2024 and will last until 01-12-2025. For each patient two years of follow-up will be collected (until a maximum of 01-12-2027). For the secondary endpoint pertaining to the sample times retrospective data will be collected from 01-02-2024 up to 01-02-2025. Remnant material will be collected in the period during the follow-up period after obtaining informed consent

#### STUDY POPULATION

#### Population (base)

The population includes adult patients (age between 18 and 70) with treatment resistant schizophrenia of schizoaffective disorder, treated with oral, once or twice-daily clozapine.

Data will be collected from mental healthcare organization GGZ-NHN. All the patients have been treated with clozapine as part of standard care, as well as sampled routinely as part of

376 standard care.

370

371

377378

379

380 381

382

383 384

385

386 387

388

389

390

391

392

393

394

#### Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria and provide informed consent. These criteria are partially based on covariates used the model by Beex et al., as it will be used in this study (22):

- Standard treatment of a stable, oral dose of clozapine for at least one week (at steady state).
- Age between 18-70 years.
- Registered time of intake as well as sampling time and dosage.
- Registered smoking status (yes/no).
- At least two samples in the elimination phase of clozapine with both clozapine and norclozapine measured.
- Measurement of the white cell count at least every three months or more often.
- Routine metabolic screening performed at moment of inclusion
- Subjects should be able to understand the study information and procedures and give informed consent or when incapacitated subjects are not reliably able to give informed consent their legal representatives should give informed consent under the condition that these subjects are willing to participate.

395 396 397

398

399

400

401

402 403

404

405

406

407 408

409 410

411

412

413

#### **Exclusion criteria**

A potential subject or specific samples that meet any of the following criteria will be excluded from this study:

- Pregnancy.
- Malignancy or treatment with immunosuppressive medication.
- Samples where cessation, start or dose change of interacting co-medication (such as valproic acid, gemfibrozil, fluvoxamine, omeprazole and cyclic oral contraceptives [21 on, 7 days off]) or changes in use of tobacco containing products occurred within seven days prior to blood sampling (21, 28, 34, 35).
- Acute inflammation, infection or samples shortly after intoxication. In case this
  information is unknown, it may be derived by large unexpected change in levels
  compared to previous or target levels.
- Not sampled at Starlet (blood collection site) or sampled by dried blood spot
- Unknown status of smoking (including vaping).
- Unknown time of intake of clozapine.
- Unknown time of blood sampling.
- If informed consent is not obtained by the patient or by a legal representative in a mentally incapacitated patient, i.e. a legally incompetent adult.

414 415 416

417

418 419

420

421 422

423

#### Sample size calculation

No calculation was performed since the effect of clozapine on the increase of metabolic markers is unknown. A rule of thumb with pharmacokinetic studies is an amount of 30 patients, however with the combination of pharmacokinetics and pharmacodynamics the variability in the endpoint will increase. Based on a previous PK/PD study which studied the relationship of the drug adalimumab with the PASI-score, a population of approximately 60 patients was sufficient for establishing a correlation with the pharmacokinetics of adalimumab

| 424<br>425<br>426<br>427 | and the clinical response measured by the PASI (36). For the secondary endpoint investigating the effect a minimum of 30 patients with 90-120 samples is likely sufficient. |
|---|---|
| 428 | TREATMENT OF SUBJECTS |
| 429<br>430 | This chapter is not applicable as this is a non-interventional study. |
| 431 | INVESTIGATIONAL PRODUCT |
| 432 | This chapter is not applicable as this is a non-interventional, retrospective study that involves |
| 433 | standard care. |
| 434 | |
| 435 | NON-INVESTIGATIONAL PRODUCT |
| 436 | This chapter is not applicable as this is a non-interventional, retrospective study that involves |
| 437 | standard care. |
| 438 | |

#### **METHODS**

#### Study parameters/endpoints

#### Main study parameter/endpoint

Correlation between serum level HbA1c and (nor)clozapine concentrations and ratio will be assessed using a PK-PD turn over model.

#### Secondary study parameters/endpoints

 The predictive performance of the model by Beex et al. (22) for our population will be assessed through calculations of the prediction error for each observation as well as the root mean square error to measure the overall prediction accuracy.

In order to study the main study point, the model by Beex et al. will have to be validated for our population first. However, since this is not the primary objective, it is noted as a secondary objective that will be performed before researching the primary endpoint. The cutoff value for the mean and median values of prediction errors is also based on clinical practice as well as the study by Veerman et al. (37) and thus set at 20%.

 Percentage difference in clozapine and norclozapine median concentrations predicted 10, 11, 13 and 14-hour post intake (based on clinical samples) compared to median concentrations at current reference sampling time of 12-hour post intake.

Based on the study of Veerman et al. an increase of 100  $\mu$ g/L is regarded as clinically relevant (37). However, measurement errors may also impact the differences between concentrations and are expressed in a percentage. Therefore, clinically relevant differences will be expressed as a percentage as well. The increase of 100  $\mu$ g/L is set off against the therapeutic window of 350-700  $\mu$ g/L up to the alert level of 1000  $\mu$ g/L. As the midpoint of this range would be 525  $\mu$ g/L, 100  $\mu$ g/L would correspond with a difference of 20%. This difference is defined as clinically relevant for this study, according to which concentrations would no longer be deemed similar and thus corresponding to the same time window or an adequate sampling time or window.

• Percentage difference in clozapine and norclozapine concentrations based on different sampling times across entire concentration-time profiles to identify optimal sampling time or window within current therapeutic window of 350-700 µg/L.

To identify the optimal sampling time or window, expected concentration-time profiles will be constructed on basis of individual PK parameters obtained by Bayesian analysis. In these profiles sampling times during which the concentration will be within the therapeutic window of 350-700  $\mu$ g/L will be identified. These graphical 'reference ranges' could point to an optimal sampling time or window. In order for a sampling time window to be found, concentrations within that window would have to be deemed similar. As a percentage difference of 20% between concentrations will be regarded as clinically relevant, concentrations within the same window are allowed a difference up to 20%. As such, a new sampling time or window might be found instead of the current window of 10 to 14 hours post intake.

- Effect of covariates on the pharmacokinetics of clozapine, the metabolite norclozapine (and CZ/NCZ ratio). Covariates to be studied include: age, estradiol, comedication (e.g. fluvoxamine), ethnicity, pharmacogenetics, smoking behaviour, inflammation markers, phenylalanine and tyrosine.
- Correlation between other metabolic parameters (such as fasting glucose, insulin, HOMA-IR, triglycerides, HDL, LDL, total cholesterol, BMI, abdominal circumference, blood pressure and heart rate), ANC and TWC, GASS-C, BSFS and PANSS-6

| 493<br>494 | regarding severity of schizophrenia and the (nor)clozapine concentrations and ratio will be assessed using a PK-PD turn over model. |
|---|---|
| | will be assessed using a FN-FD turn over model. |
| 495 | The effect of certical concentration and genetics on the correlation of (nor)eleganine |
| 496 | <ul> <li>The effect of cortisol concentration and genetics on the correlation of (nor)clozapine<br/>concentrations and/or ratio on the metabolic markers</li> </ul> |
| 497 | concentrations and/or ratio on the metabolic markers |
| 498 | |
| 499 | Other study neversators |
| 500<br>501 | Other study parameters Demographics |
| 502 | - Sex (male/female). |
| 503 | · |
| | - Age (year). |
| 504 | - Estradiol indirectly (premenopausal/postmenopausal female / male). |
| 505 | - Ethnicity (Caucasian/African-Caribbean/Asian/other). |
| 506 | Climical maramatara |
| 507 | Clinical parameters |
| 508 | - Indication for clozapine use (diagnosis treatment resistant schizophrenia or schizoaffective |
| 509 | disorder). |
| 510 | - Duration of illness. |
| 511 | - Duration of clozapine treatment. |
| 512 | - Dosage scheme. |
| 513 | - Baseline PANSS-6, regarding severity of schizophrenia |
| 514 | Oth on a grant atoms |
| 515 | Other parameters Tabagas amplified behaviour (vac/pa, including amount (prespectively)) and vaning |
| 516 | - Tobacco smoking behaviour (yes/no, including amount (prospectively)) and vaping |
| 517 | (yes/no). |
| 518 | - Interacting co-medication such as strong CYP3A4-inductors (gemfibrozil, apalutamide, |
| 519 | carbamazepine, efavirenz, enzalutamide, phenobarbital, phenytoin, St. John's wort, |
| 520 | lumacaftor, mitotane, nevirapine, primidone, rifabutin, rifampicin) or level increasing drugs |
| 521 | such as fluvoxamine, fluoxetine or sertraline, CYP1A2 inhibitors such as ciprofloxacin, or |
| 522 | inductors such as omeprazole, oral contraceptives and valproic acid). |
| 523 | - Gemfibrozil and valproic acid use, as both inhibit renal clearance of norclozapine (38). |
| 524<br>525 | - Patient specific target level if this falls outside of the therapeutic window of 350-700 μg/L, in |
| 525 | order to be able to identify these levels as expected normal target levels instead of toxic or |
| 526 | caused by (in)adherence, interactions or infection Reason for blood collection if available (routine or otherwise: possible toxicity, infection, |
| 527 | CRP and BSE if recently measured and known, change in dosage or co-medication). |
| 528<br>529 | CRF and BSE in recently measured and known, change in dosage or co-medication). |
| 530 | |
| 531 | Randomisation, blinding and treatment allocation |
| 532 | Not applicable |
| 533 | Study procedures |
| 534 | Not applicable, patients will not undergo any (additional) procedures for research |
| 535 | purposes. All samples will be taken as part of standard care for treatment purposes. |
| 536 | Withdrawal of individual subjects |
| 537 | Not applicable |
| 538 | Specific criteria for withdrawal (if applicable) |
| 539 | Not applicable |
| 540 | Replacement of individual subjects after withdrawal |
| 541 | Not applicable |
| 542 | Follow-up of subjects withdrawn from treatment |
| 543 | Not applicable |
| 544 | Premature termination of the study |
| 545 | Not applicable |
| | • • |

# 547 **SAFETY REPORTING**

This chapter is not applicable as this is a non-interventional, retrospective study that involves standard care.

549 550

548

Version number: 2, 22-11-2024 19 of 28

#### STATISTICAL ANALYSIS

# 

# 

# 

# Primary study parameter(s)

PK analyses will be performed using nonlinear-mixed-effects modelling (NONMEM) software (version 7.4.2, ICON Development Solution, Gaithersburg, MD, USA). Software like R (www.rproject.org), Pirana and Xpose (version 4.3.2, Niclas Jonsson and Mats Karlsson, Uppsala, Sweden) will be used for graphical display and evaluation of the models (including goodness of fit plots).

Previously Beex et al., while studying the comparability of pharmacokinetics of clozapine and norclozapine with once- and twice-daily dosing, developed a population PK model using NONMEM (13). Furthermore, their popPK model has incorporated patient-specific covariate smoking to further refine pharmacokinetic parameter estimates and improve the accuracy of dosing. Their base model describes clozapine by a two-compartment model with a transit compartment describing the delay in absorption and linear elimination consisting of combined excretion and formation of the metabolite norclozapine. This model was extended with a one-compartment model for norclozapine with first-order elimination (Figure 2, excerpt from their study).



Figure 2. Schematic representation of the structural model.

AMT = amount, CI = clearance of clozapine, CI2 = clearance of norclozapine, CLZ = clozapine, FMET = fraction metabolised, ktr = transit compartment rate constant, NCLZ = norclozapine, Q = intercompartimental clearance

Their final model tested for several covariates: total body weight, BMI, age, sex, AGP concentrations, albumin concentrations, CRP, and smoking status. Only smoking had a significant effect on clozapine clearance (not on norclozapine clearance). Based on this model, clearance of clozapine is 55% higher in smokers than in non-smokers. Table 2 is an excerpt of the overview of parameter estimates of both base and final model.

**Table 2.** Overview of parameter estimates of base model, final model and SIR. SIR was run on 2000 samples and 1000 resamples. CI = confidence interval, CLZ = clozapine, CI/F = apparent clearance of clozapine, CI/F'= apparent clearance of norclozapine, FMET = fraction of clozapine metabolised into norclozapine, Ktr = transit rate constant, Q = intercompartimental clearance, OFV = objection function value, NCLZ = norclozapine, RSE = relative standard error, SIR = sampling importance resampling, Vcentral / F= apparent central volume of distribution of clozapine, Vperipheral / F= apparent peripheral volume of distribution of clozapine, V/ F' = apparent volume of distribution of norclozapine. FIX = fixed value

| Parameter | Base model (RSI | %) Final model (RSE | %) SIR (95% CI) |
|---|---|---|---|
| CI/F CLZ (L/h) | 30.8 (7.4%) | 22.2 (14.8%) | 22.2 (18.0 - 28.0) |
| Smoking on CI/F | - | 1.55 (16.4%) | 1.55 (1.20 - 1.96) |
| V <sub>central</sub> /F CLZ (L) | 328 (11.4%) | 328 (11.3%) | 328 (257 - 422) |
| V <sub>peripheral</sub> /F CLZ (L) | 285 (17.1%) | 286 (17.0%) | 286 (199 - 394) |
| Q (L/h) | 86.0 (22.3%) | 86.0 (21.9%) | 86.0 (60.1 - 130.1) |
| Ktr (h-1) | 1.23 (10.0%) | 1.23 (10.0%) | 1.23 (0.99 - 1.52) |
| CI/F' NCLZ (L/h) | 36.1 (8.0%) | 36.1 (8.0%) | 36.1 (31.3 - 41.7) |
| V/F' NCLZ (L) | 746 (72.0%) | 751 (72.2%) | 751 (418 - 1796) |
| FMET | 0.66 FIX | 0.66 FIX | 0.66 FIX |
| Interindividual varial | bility (%) | | |
| IIV CI/F CLZ | 49.7 (8.6%) | 45.1 (10.0%) | 43.0 (36.7 - 53.4) |
| IIV V <sub>central</sub> /F | 63.7 (10.9%) | 63.5 (12.4%) | 58.2 (44.4 - 72.9) |
| IIV V <sub>peripheral</sub> / F CLZ | 72.8 (28.9%) | 72.7 (29.0%) | 62.8 (46.8 - 84.6) |
| IIV Ktr | 69.6 (16.6%) | 69.6 (16.5%) | 50.0 (42.1 - 59.4) |
| IIV CI/F' NCLZ | 53.3 (8.6%) | 53.3 (8.9%) | 65.1 (29.7 - 104.3) |
| Proportional error<br>CLZ (%) | 13.2 (9.1%) | 13.2 (9.1%) | 13.2 (12.0 - 14.7) |
| Proportional error<br>NCLZ (%) | 18.3 (8.3%) | 18.3 (8.2%) | 18.2 (16.7 – 20.0) |
| OFV (-2 LL) | 7610.26 | 7602.50 (-7.76) | |

Subsequently, their developed final population PK model will be used to predict concentration-time profiles for clozapine and norclozapine under various dosages and sampling schedules on basis of individual PK parameters obtained by Bayesian analysis. Collected data will be inserted into R as well as relevant patient-specific demographic, clinical and laboratory data. A new database suitable for PK analyses of clozapine will be constructed in NONMEM. In order to do this the clozapine dose, measured concentration data along with time of intake and sampling time will be taken into account. Subsequently, PK profiles will be predicted. The reference window to be targeted will be 350-700  $\mu$ g/L for clozapine. Deviation from this window will be allowed for patients who, according to their psychiatrist or nurse specialist or other practitioner, have a higher or lower target level than the defined therapeutic window with good therapeutic effect. This will only be allowed based on the psychiatrist/nurse specialist/practitioner's information and help identify these levels as expected normal target levels instead of toxic or caused by inadherence, interactions or infection.

 The first step before researching the primary endpoint, is the performance of an external validation (see secondary study parameter(s) below). Afterwards, the current study population will be studied in order to research the primary endpoint. To analyse this, the concentration-time data will be used to develop PK/PD turn-over models to estimate the parameters (Kin, Kout, Emax and EC50) linking the pharmacokinetics of clozapine and norclozapine to HbA1c serum levels. Once the structural PK/PD model is developed, the between subject variability and residual unexplained variability of the estimated pharmacokinetic parameters will be assessed.

 A univariate covariate analysis will be performed to check for associations between the patient-related factors on parameters of the PD model using a  $\chi 2$  test-statistic. Covariates with a significant association in the univariate analysis will be included in the multivariate analysis. Covariates that remain significant in the multivariate analysis will be included in the final pharmacodynamic model. This final model will be validated using visual predictive check (VPC's) and using a bootstrap procedure the robustness of the model will be tested. The latter two procedures will be performed using Piraña and Pearl speaks NONMEM (PsN) software.

#### Secondary study parameter(s)

For the external validation of the model, predicted profiles will be compared to the observed data of our population (which is regarded as an external data set). Prediction error (PE) for each predicted concentration (PE) was defined through the following equation:

$$ext{PE}_i = rac{ ext{(Observed}_i - ext{Predicted}_i)}{ ext{Observed}_i} imes 100$$

 where Observed<sub>i</sub> and Predicted<sub>i</sub> represent the *i*th observed and predicted concentrations, respectively. The root mean square error (RMSE) prediction error was also calculated using the following equation:

$$RMSE = \sqrt{\frac{1}{n} \sum_{i=1}^{n} (Observed_i - Predicted_i)^2}$$

where n represents the total number of concentrations. A population PK model was regarded as valid for our clinical settings when both the mean and median values of PE were less than 20%. As stated earlier, the external validation of the model by Beex et al. will be performed before researching our primary goal.

 Based on the predicted concentration-time profile for all participants, the percentage difference in predicted clozapine and norclozapine concentrations between different sampling times will be calculated. The 12-h time point will be set as reference and compared to concentrations predicted (or measured if available) at 10, 11, 13 and 14 hours-post intake concentrations. Plasma concentrations taken at steady state should be comparable to others within an acceptable time window. As stated earlier, concentrations are regarded as comparable if the total percentage difference does not exceed 20%. This includes expected bias and imprecision in measurement and interoccassion and interindividual variability. This difference is defined as clinically relevant for this study, according to which concentrations would no longer be deemed similar and thus corresponding to the same time window or an adequate sampling time or window.

 Statistical significance will be tested through generalized linear mixed models for proportions, in which the proportion of clinically relevant differences per time point versus t=12 will be compared. For descriptive statistics, continuous outcomes are presented as medians and ranges between minimum and maximum values with corresponding confidence intervals, when applicable. Categorical outcomes are reported as numbers and proportions (n (%)). Two tailed p-values of < 0.05 based on  $\chi 2$  with one degree of freedom were considered statistically significant.

Based on the clinical patient data, predicted concentration-time profiles, averaged for each subject, will be portrayed for different oral dosages. The (new) optimal sampling window will be based on the time window during which the difference in measured clozapine and

norclozapine concentrations in the predicted profile is smaller than 20% as well as within the defined therapeutic window of  $350\text{-}700~\mu\text{g/L}$  for clozapine. If needed, deviation from this window will be allowed for patients with different target levels as described before. This will be only be allowed based on the psychiatrist/nurse specialist/practitioner's information. If a window cannot be found, then sampling times will be noted during which clozapine concentrations fall within the defined therapeutic window. The student's t-test for paired data was used to analyse differences in median serum concentrations across sampling times.

Aside from the metabolic parameters mentioned in the primary endpoint, correlation with other metabolic parameters (such as fasting glucose, insulin, HOMA-IR, triglycerides, HDL, LDL, total cholesterol, BMI, abdominal circumference, blood pressure and heart rate), ANC, TWC. GASS-C and BSFS with the concentrations will be studied. The concentration-time data will be used to develop PK/PD turn-over models to estimate the parameters (Kin, Kout, Emax and EC50) linking the pharmacokinetics of clozapine and norclozapine to these parameters. Once the structural PK/PD model is developed, the between subject variability and residual unexplained variability of the estimated pharmacokinetic parameters will be assessed. A univariate covariate analysis will be performed to check for associations between the patient-related factors on parameters of the PD model using a  $\chi 2$  test-statistic. Covariates with a significant association in the univariate analysis will be included in the multivariate analysis. Covariates that remain significant in the multivariate analysis will be included in the final pharmacodynamic model. This final model will be validated using visual predictive check (VPC's) and using a bootstrap procedure the robustness of the model will be tested. The latter two procedures will be performed using Piraña and Pearl speaks NONMEM (PsN) software.

Using an univariate analysis in NONMEM the association of patient-related factors on the pharmacokinetic parameters of clozapine will be tested using a  $\chi 2$  test-statistic. The covariates that will be included in the univariate analysis include age, gender, premenopauzal/postmenopausal female/male, ethnicity, weight, height, CRP, BSE, smoking behaviour, comedication with fluvoxamine (dosage) and genotypes. Covariates with a significant association in the univariate analysis will be included in the multivariate analysis. Covariates that remain significant in the multivariate analysis will be included in the final pharmacokinetic model. This final model will be validated using visual predictive check (VPC's) and using a bootstrap procedure the robustness of the model will be tested. The latter two procedures will be performed using Piraña and Pearl speaks NONMEM (PsN) software. The final pharmacokinetic model will then be used to create concentration-time curves for each individual participating in the PK/PD study.

#### Other study parameters

Baseline characteristics will be depicted by means of summary statistics: mean  $\pm$  SD for normally distributed continuous variables and median  $\pm$  interquartile range for non-normally distributed continuous variables. Proportions will be calculated for categorical variables.

# Interim analysis (if applicable)

698 Not applicable.

#### ETHICAL CONSIDERATIONS 699 This is an observational cohort study in which the data will be collected retrospectively. The 700 subjects included in this study will not undergo any additional procedures. After gaining 701 702 permission by the Advisory Committee on Local Feasibility of the GGZ-NHN, all subjects will be asked informed consent before participation. Informed consent will be asked in 703 704 accordance with the General Data Protection Regulation (GDPR). Their Electronic Health Record (EHR) will be viewed by the treating psychiatrist, physician, nurse specialist, or other 705 706 doctor/practitioner. Data collected by the practitioner will be used for the dataset. 707 Additionally, information such as plasma levels is collected through Labosys rapports for which informed consent is given according to standard procedure for blood collection. 708 Remnant material from laboratory procedures performed as part of routine clinical care will 709 710 be collected and stored. 711 712 **Regulation statement** This research will be conducted in accordance with Good clinical practice (GCP) and GDPR. 713 714 715 **Recruitment and consent** 716 This study will be submitted to the local review committee of the GGZ-NHN. Letter and informed consent are attached as separate documents. 717 718 Objection by minors or incapacitated subjects (if applicable) 719 720 Not applicable. Benefits and risks assessment, group relatedness 721 722 Not applicable. 723 Compensation for injury 724 Not applicable. Incentives (if applicable) 725 Not applicable. 726 727

Data regarding sex, age, plasma levels of both clozapine and norclozapine, time of intake

# ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION Handling and storage of data and documents

730

731732733

and sampling time will be collected through reports from Labosys (Alkmaar). This data is sourced from the blood collection site, where requesting psychiatrists, physicians, nurse specialists, or other doctors/practitioners are required to fill in this information. All specified laboratory parameters (see above) from both GGZ-NHN and other sources of requests for laboratory diagnostic procedures (i.e. general practitioner, specialist internal medicine) within the period of follow-up will be used for analysis. Time of intake will be collected from the patients before the sampling time at the collection site (Starlet) according to standard practice. Due to new ISO regulations, there are upcoming changes in standard practice for blood collection at the main site. These changes will require requesting doctors to fill in more information at every blood collection request such as: smoking (yes/no), dosage, reason for blood collection (routine or otherwise: possible toxicity, infection, change in dosage). Once these changes have followed through, this data can also be collected through Labosys. Comedication will be retrieved through the patient's public pharmacy.

746747748

749

750 751

752

753 754

755

756 757

758

759

760

761

762

763

764 765

766

767

740

741

742

743744

745

Before implementation of these changes, information on smoking, dosage and reason for blood collection will be collected through the treating psychiatrist/nurse specialist/practitioner who has access to the patient's electronic health record if needed. Other information to be gathered by the treating psychiatrist/nurse specialist/practitioner includes: weight and BMI, ethnicity, diagnosis (of schizophrenia or other psychiatric disorder), pregnancy, interacting co-medication (including newly started, stopped medication and changes in dosages within a week of sampling time). Data regarding metabolic parameters such as fasting glucose, serum level HbA1c, triglycerides, HDL, LDL, total cholesterol, abdominal circumference, BMI and blood pressure and heart rate will be collected through reports through Nexus and mConsole (Alkmaar), as well as the absolute neutrophil count (ANC) and the outcomes of the Bristol Stool Form Scale (BSS) assessment, the Glasgow Antipsychotic Side-effect Scale for Clozapine (GASS-C) questionnaire and the Positive and Negative Syndrome Scale (PANSS-6) questionnaire will be collected through Nexus and mConsole (Alkmaar). Clinical data needed from the dedicated includers (co-investigators, with an affiliation to the GGZ-NHN) will be collected through a simple case report form. This information will be collected at the moment of inclusion and at the end of the study (retrospectively) in case any changes occur during the study period. Biologic material collected as part of laboratory investigation as part of routine clinical care after obtaining informed consent will be stored at the laboratories of the North West Clinics until all laboratory procedures pertaining the investigation are completed (metabolic enzymes, the genes CYP2C19 and CYP3A4 and genes related to metabolic markers).

768 769 770

771

772773

Missing data (unless described in the inclusion or exclusion criteria) will be allowed. Native speakers, if available, will be asked to deduct a patient's ethnicity based on their name in case the ethnicity is unknown before regarding this as missing data. If data, such as BMI or CRP, are not reported in the patient's medical file the event will be recorded as 'missing data' or as not occurred.

774775776

777

778 779 During the study period, data collected from the psychiatrist/nurse specialist/practitioner/dedicated includer will be linked to data collected from Labosys according to date of birth and name. Patient data will be encoded. The key will be safeguarded by the coordinating investigator and principal investigators. Furthermore collected data will be stored for 15 years.

780 781 782

783

The results, discussion and conclusion of the study will be reported and shared in an abstract, manuscript and registration presentation in accordance to the principles of the

| 784<br>785<br>786<br>787 | ICMJE guidelines. Information concerning this study's processes and data is confidential and its rights belong to GGZ-NHN, NWZ Alkmaar and Amsterdam UMC. |
|---|---|
| 788 | Monitoring and Quality Assurance |
| 789 | Not applicable |
| 790 | Amendments |
| 791 | Not applicable |
| 792 | Annual progress report |
| 793 | Not applicable |
| 794 | Temporary halt and (prematurely) end of study report |
| 795 | Not applicable |
| 796 | Public disclosure and publication policy |
| 797 | Not applicable |
| 798 | |
| 799 | STRUCTURED RISK ANALYSIS |
| 800 | Not applicable |
| 801 | |
| 802 | |

#### **REFERENCES**

807

811

812

813

814

815

822

823 824

825

826

827

828

829

830

834

835

- 1. Hiemke C, Bergemann N, Clement HW, Conca A, Deckert J, Domschke K, et al. Consensus Guidelines for Therapeutic Drug Monitoring in Neuropsychopharmacology: Update 2017. Pharmacopsychiatry. 2018;51(1-02):9-62.
- Hiemke C, Baumann P, Bergemann N, Conca A, Dietmaier O, Egberts K, et al. AGNP
   Consensus Guidelines for Therapeutic Drug Monitoring in Psychiatry: Update 2011.
   Pharmacopsychiatry. 2011:44(6):195-235.
  - 3. Schoretsanitis G, Kane JM, Correll CU, Marder SR, Citrome L, Newcomer JW, et al. Blood Levels to Optimize Antipsychotic Treatment in Clinical Practice: A Joint Consensus Statement of the American Society of Clinical Psychopharmacology and the Therapeutic Drug Monitoring Task Force of the Arbeitsgemeinschaft für Neuropsychopharmakologie und Pharmakopsychiatrie. J Clin Psychiatry. 2020;81(3).
- 4. Schulte PFJ BB, Bogers J, Cohen D, van Dijk D. . Guideline for the use of clozapine; explanatory supplement accompanying a guideline. <a href="http://www.clozapinepluswerkgroep.nl/wp-content/uploads/2013/07/Guideline-for-the-useof-Clozapine-2013.pdf">http://www.clozapinepluswerkgroep.nl/wp-content/uploads/2013/07/Guideline-for-the-useof-Clozapine-2013.pdf</a>. [updated Updated 2013. Accessed February 2nd, 2024].
- 5. Yuen JWY, Kim DD, Procyshyn RM, Panenka WJ, Honer WG, Barr AM. A Focused Review of the Metabolic Side-Effects of Clozapine. Front Endocrinol (Lausanne). 2021;12:609240.
  - 6. Li XH, Zhong XM, Lu L, Zheng W, Wang SB, Rao WW, et al. The prevalence of agranulocytosis and related death in clozapine-treated patients: a comprehensive meta-analysis of observational studies. Psychol Med. 2020;50(4):583-94.
    - 7. Costa-Dookhan KA, Agarwal SM, Chintoh A, Tran VN, Stogios N, Ebdrup BH, et al. The clozapine to norclozapine ratio: a narrative review of the clinical utility to minimize metabolic risk and enhance clozapine efficacy. Expert Opin Drug Saf. 2020;19(1):43-57.
    - 8. Jessurun NT, Derijks HJ, van Marum RJ, Jongkind A, Giraud EL, van Puijenbroek EP, Grootens KP. Body weight gain in clozapine-treated patients: Is norclozapine the culprit? Br J Clin Pharmacol. 2022;88(2):853-7.
- 9. Park R, Kim S, Kim E. Relationship of Change in Plasma Clozapine/N-desmethylclozapine Ratio with Cognitive Performance in Patients with Schizophrenia. Psychiatry Investig. 2020;17(11):1158-65.
  - 10. Schoretsanitis G, Kane JM, Ruan CJ, Spina E, Hiemke C, de Leon J. A comprehensive review of the clinical utility of and a combined analysis of the clozapine/norclozapine ratio in therapeutic drug monitoring for adult patients. Expert Rev Clin Pharmacol. 2019;12(7):603-21.
- Yuen JWY, Wu C, Wang CK, Kim DD, Procyshyn RM, Honer WG, Barr AM. A comparison of
   the effects of clozapine and its metabolite norclozapine on metabolic dysregulation in rodent models.
   Neuropharmacology. 2020;175:107717.
- Tan MSA, Honarparvar F, Falconer JR, Parekh HS, Pandey P, Siskind DJ. A systematic review and meta-analysis of the association between clozapine and norclozapine serum levels and peripheral adverse drug reactions. Psychopharmacology (Berl). 2021;238(3):615-37.
- Lu ML, Lane HY, Lin SK, Chen KP, Chang WH. Adjunctive fluvoxamine inhibits clozapine-related weight gain and metabolic disturbances. J Clin Psychiatry. 2004;65(6):766-71.
- Lu ML, Chen TT, Kuo PH, Hsu CC, Chen CH. Effects of adjunctive fluvoxamine on metabolic
   parameters and psychopathology in clozapine-treated patients with schizophrenia: A 12-week,
   randomized, double-blind, placebo-controlled study. Schizophr Res. 2018;193:126-33.
- Polcwiartek C, Nielsen J. The clinical potentials of adjunctive fluvoxamine to clozapine treatment: a systematic review. Psychopharmacology (Berl). 2016;233(5):741-50.
- Willcocks IR, Legge SE, Nalmpanti M, Mazzeo L, King A, Jansen J, et al. Clozapine
   Metabolism is Associated With Absolute Neutrophil Count in Individuals With Treatment-Resistant
   Schizophrenia. Front Pharmacol. 2021;12:658734.
- 17. Okhuijsen-Pfeifer C, Cohen D, Bogers J, de Vos CMH, Huijsman EAH, Kahn RS, Luykx JJ. Differences between physicians' and nurse practitioners' viewpoints on reasons for clozapine underprescription. Brain Behav. 2019;9(7):e01318.
- 856 18. Spina E, Avenoso A, Facciolà G, Scordo MG, Ancione M, Madia AG, et al. Relationship 857 between plasma concentrations of clozapine and norclozapine and therapeutic response in patients 858 with schizophrenia resistant to conventional neuroleptics. Psychopharmacology (Berl). 859 2000;148(1):83-9.
- Kronig MH, Munne RA, Szymanski S, Safferman AZ, Pollack S, Cooper T, et al. Plasma clozapine levels and clinical response for treatment-refractory schizophrenic patients. Am J Psychiatry. 1995;152(2):179-82.

- 863 20. Jakobsen MI, Larsen JR, Svensson CK, Johansen SS, Linnet K, Nielsen J, Fink-Jensen A.
- 864 The significance of sampling time in therapeutic drug monitoring of clozapine. Acta Psychiatr Scand.
- 865 2017;135(2):159-69.
- 866 Mylan. Summary of Product Characteristics - UK Clozaril 25 mg tablets [updated 12-05-21.
- 867 2020].
- 868 Beex-Oosterhuis MM, Lau C, Verloop S, Grootens KP, Faber G, Gool vAR, et al. The impact
- 869 of once-daily dosing on the pharmacokinetics of clozapine and norclozapine. Unpublished, PhD thesis. 870 2023.
- 871 23. VanderZwaag C, McGee M, McEvoy JP, Freudenreich O, Wilson WH, Cooper TB. Response 872 of patients with treatment-refractory schizophrenia to clozapine within three serum level ranges. Am J 873 Psychiatry. 1996;153(12):1579-84.
- 874 Procyshyn RM, Vila-Rodriguez F, Honer WG, Barr AM. Clozapine administered once versus 875 twice daily: does it make a difference? Med Hypotheses. 2014;82(2):225-8.
- 876 Kitagawa K, So R, Nomura N, Tsukahara M, Misawa F, Kodama M, et al. Clozapine Once-
- Daily Versus Divided Dosing Regimen: A Cross-sectional Study in Japan. J Clin Psychopharmacol. 877 878 2022;42(2):163-8.
- 879 Moscou TV, SRT. Clozapine/norclozapine plasma level ratio and cognitive functioning in
- 880 patients with schizophrenia spectrum disorders: a systematic review. Therapeutic Advances in 881 Psychopharmacology, 2024; Accepted.
- 882 Pu X, Gao Y, Li R, Li W, Tian Y, Zhang Z, Xu F. Biomarker Discovery for Cytochrome P450 883 1A2 Activity Assessment in Rats, Based on Metabolomics. Metabolites. 2019;9(4).
- 884 Geers LM, Cohen D, Wehkamp LM, van Wattum HJ, Kosterink JGW, Loonen AJM, Touw DJ.
- 885 Population pharmacokinetic model and limited sampling strategy for clozapine using plasma and dried 886 blood spot samples. Ther Adv Psychopharmacol. 2022;12:20451253211065857.
- 887 Perera V, Bies RR, Mo G, Dolton MJ, Carr VJ, McLachlan AJ, et al. Optimal sampling of
- antipsychotic medicines: a pharmacometric approach for clinical practice. Br J Clin Pharmacol. 888
- 2014;78(4):800-14. 889
- 890 Shang DW, Li LJ, Wang XP, Wen YG, Ren YP, Guo W, et al. Population
- 891 pharmacokinetic/pharmacodynamic model of clozapine for characterizing the relationship between
- 892 accumulated exposure and PANSS scores in patients with schizophrenia. Ther Drug Monit.
- 893 2014;36(3):378-86.
- 894 31. Wester VL, Koper JW, van den Akker EL, Franco OH, Stolk RP, van Rossum EF.
- 895 Glucocorticoid receptor haplotype and metabolic syndrome: the Lifelines cohort study. Eur J 896 Endocrinol. 2016;175(6):645-51.
- van Walree ES, Jansen IE, Bell NY, Savage JE, de Leeuw C, Nieuwdorp M, et al. 897
- 898 Disentangling Genetic Risks for Metabolic Syndrome. Diabetes. 2022;71(11):2447-57.
- 899 Hynes C, Keating D, McWilliams S, Madigan K, Kinsella A, Maidment I, et al. Glasgow
- 900 Antipsychotic Side-effects Scale for Clozapine - Development and validation of a clozapine-specific 901 side-effects scale. Schizophr Res. 2015;168(1-2):505-13.
- 902 Reeves S, Bertrand J, Obee SJ, Hunter S, Howard R, Flanagan RJ. A population
- 903 pharmacokinetic model to guide clozapine dose selection, based on age, sex, ethnicity, body weight 904 and smoking status. Br J Clin Pharmacol. 2024;90(1):135-45.
- 905 Barclay J, McCollum B, Schoretsanitis G, de Leon J. Gemfibrozil May Decrease Norclozapine 906 Elimination: A Case Report. J Clin Psychopharmacol. 2019;39(4):405-7.
- 907 van Huizen A, Bank P, van der Kraaij G, Musters A, Busard C, Menting S, et al. Quantifying 908 the Effect of Methotrexate on Adalimumab Response in Psoriasis by Pharmacokinetic-
- Pharmacodynamic Modeling. J Invest Dermatol. 2024;144(4):794-801.e6. 909
- 910 Veerman SRT, Moscou T, Bogers J, Cohen D, Schulte PFJ. Clozapine and COVID-19
- 911 Vaccination: Effects on blood levels and leukocytes. An observational cohort study. Acta Psychiatr
- 912 Scand. 2022;146(2):168-78.

- van Weringh G, van Koolwijk L, de Haan L, Touw DJ, de Koning MB. Paralytic ileus in a 913
- 914 patient on clozapine therapy showing an inverted clozapine/norclozapine ratio after switching valproic
- 915 acid to carbamazepine; a case report. Ther Adv Psychopharmacol. 2024;14:20451253241255487.

Version number: 2, 22-11-2024